CLINICAL TRIAL: NCT06549062
Title: Pharmacokinetics and Pharmacodynamics of Intravenous Paracetamol/Acetaminophen in Morbidly Obese and Non- Obese Patients.
Brief Title: Pharmacokinetics and Pharmacodynamics of Intravenous Paracetamol in Morbidly Obese and Non- Obese Patients.
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Patrick F Wouters, MD PhD, head of department, University Hospital, Ghent
Other Study IDs: BC-07469
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Acetaminophen Toxicity; Obesity, Morbid
Keywords: acetaminophen pharmacokinetics; obesity; NAPQI protein adducts; CYP 2E1
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples with simultaneous synchronised capillary blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese patients WHO class > 2: patients with a BMI > 35 undergoing laparoscopic surgery. venous and capillary blood samples are collected to determine the concentrations of acetaminophen and its metabolites after intravenous administration of a first dose of 2g acetaminophen and after a fifth dose of 1g acetaminophen in steady state conditions.
- non obese and overweight patients: patients with a BMI between 18,5 - 30 undergoing laparoscopic surgery. Venous and capillary blood samples are collected to determine the concentrations of acetaminophen and its metabolites after intravenous administration of a first dose of 2g acetaminophen and after a fifth dose of 1g acetaminophen in steady state conditions.

SUMMARY:
Obese patients may need higher doses of acetaminophen (APAP) for adequate analgesia, due to increased total clearance and distribution volume. APAP-induced hepatotoxicity is mainly caused through CYP2E1 pathway. Its activity is induced by obesity, potentially endangering the safety profile of APAP. Metabolic-dysfunction associated liver disease (MASLD) is an important associated risk factor for APAP induced-hepatotoxicity.

The primary endpoint of this study is to validate Van Rongen's prediction model on plasma concentration of paracetamol and its metabolites and extend it to the steady state phase over a period of 30 hours by measuring plasma concentrations of paracetamol and its metabolites and comparing them with the plasma concentrations predicted by the model by Van Rongen et al.

In addition, results obtained from venous blood will be compared with results obtained via VAMS after finger stick. If VAMS correlates well with plasma concentrations of paracetamol and its NAPQI adducts, future interventional studies may utilize the patient-friendly VAMS technology in an effort to further investigate the safety and efficacy of higher doses of paracetamol in obese patients and possibly other patient groups.

The secondary endpoints of this study are liver function tests before and after 30hrs of paracetamol administration, the VAS pain scores, the surgical pleth index (SPI) and the consumption of piritramide as recorded by a PCIA pump.

DETAILED DESCRIPTION:
A. Pharmacokinetics and pharmacodynamics of Intravenous Paracetamol in morbidly obese and non- obese patients.

Study design: interventional, stratified, controlled, prospective cohort trial

B. Hypothesis morbidly obese patients have increased CYP2E1-mediated oxidation of paracetamol, requiring higher dosage to achieve therapeutic concentrations. Higher CYP2E1 activity will produce more of the toxic NAPQI. The concentration of NAPQI adducts are a biomarker of potential liver toxicity. We expect to find ineffective plasma paracetamol concentrations + higher NAPQI adducts in the venous blood samples of obese patients compared to the non-obese patients, as confirmed by Volumetric absorptive microsampling (VAMS) from capillary blood. Based on our results, future studies can explore higher paracetamol dosage in obese using capillary sampling methods.

C. Background:

Paracetamol still is the cornerstone of non-opioid analgesia in the obese patient. Current dosing recommendations for acetaminophen limit the adult dose to 4g / day regardless of an obese body constitution.

Recent publications have shown that a higher dose of paracetamol may be required to achieve adequate concentrations in morbidly obese patients due to increased CYP2E1-mediated oxidation of paracetamol (Van Rongen et al. Clin Pharmacokinet. 2016).

In contrast, the increased CYP2E1 activity will also lead to production of the toxic paracetamol metabolite N-Acetyl-p-benzoquinone imine (NAPQI). NAPQI forms compounds or adducts with specific liver proteins. The concentration of NAPQI adducts correlates with the degree of liver damage and can be considered as a biomarker of potential liver toxicity.

Blood sampling is needed to assess plasma concentrations of paracetamol and the NAPQI adducts. Recently, the Volumetric Absorptive MicroSampling (VAMS) method has become available as a minimally invasive sampling strategy, requiring only 10 µl of capillary blood and has been validated for quantitative analysis of paracetamol and the NAPQI adducts in blood and CSF. (Delahaye, Dhont et al. 2019)

Specific objectives:

The primary endpoint of this study is to validate Van Rongen's prediction model on plasma concentration of paracetamol and its metabolites and extend it to the steady state phase over a period of 30 hours by measuring plasma concentrations of paracetamol and its metabolites and comparing them with the plasma concentrations predicted by the model by Van Rongen et al.

In addition, results obtained from venous blood will be compared with results obtained via VAMS after finger stick. If VAMS correlates well with plasma concentrations of paracetamol and its NAPQI adducts, future interventional studies may utilize the patient-friendly VAMS technology in an effort to further investigate the safety and efficacy of higher doses of paracetamol in obese patients and possibly other patient groups.

The secondary endpoints of this study are liver function tests before and after 30hrs of paracetamol administration, the VAS pain scores, the surgical pleth index (SPI) and the consumption of piritramide as recorded by a PCIA pump.

Methods:

The obese cohort group will consist of 40 obese patients undergoing elective laparoscopic bariatric surgery. The control group will consist of non-obese patients undergoing laparoscopic GI surgery because laparoscopic surgery can alter the metabolism of paracetamol. both study groups will be stratified to achieve an equal gender composition due to gender differences in paracetamol metabolism.

Sample size:

70 patients in total (15 male control patients, 15 female control patients, 20 morbidly obese men and 20 morbidly obese women).

Inclusion criteria for obese patients:

* BMI> 35 kg.m-2 undergoing laparoscopic surgery.
* Patients >18 years old
* ASA physical classification II to III

Inclusion criteria for control patients:

* Patients 18.5 ≤ BMI ≤ 30 kg.m-2 undergoing elective laparoscopic surgery (Nissen procedure, inguinal hernia repair, laparoscopic bowel surgery and cholecystectomy).
* ASA physical classification I to III
* Patients > 18 yrs

Exclusion criteria for obese and non-obese patients:

Renal impairment eGFR <30ml / min, Liver disease liver enzymes> 3X normal values or documented liver pathology in the medical record, Patients with Gilbert-Meulengracht syndrome, pregnancy, Chronic alcohol intake or alcohol use within the last 72 hours, Patients treated with drugs known to affect CYP2E1 and UGT (UDP-glucuronosyltransferase), Chronic malnutrition, Paracetamol allergy, Clinical study last 30 days.

Procedures:

After induction, a second intravenous catheter for blood sampling is placed in a large vein of the contralateral arm of the first intravenous line and kept patent with a positive pressure needles connector

The paracetamol dose administered is part of the "standard of care" and is not a study specific intervention. All paracetamol will be administered over 15 minutes with a volumetric pump.

T0: administration of standard paracetamol (2g) dose after induction of anesthesia, followed by IV 1g / 6hrs postoperatively up to 30 h after first administration.

In addition to paracetamol, the patients receive a IV- dose of ibuprofen (600mg every 8h) and a patient controlled intravenous analgesia pump with piritramide (1mg/ml).

Routine monitoring:

Non-invasive blood pressure (NIBP), electrocardiography (ECG), pulse oximetry (SpO2) with a Surgical Pleth Index (SPI) module (GE-Health care). The SPI index is a measure of the balance between nociception/antinociception.

The first group consists of 40 obese patients undergoing elective laparoscopic surgery. The control group consists of non-obese patients undergoing laparoscopic GI surgery because laparoscopy can alter paracetamol metabolism. Both groups will be stratified to an equal gender composition due to gender differences in paracetamol metabolism. all patients receive the same dose of paracetamol. a second intravenous catheter for blood sampling is placed in a large vein of the contralateral arm.

Liver function (AST, ALT, prothrombin time [PT], c-glutamyl transpeptidase [c-GT] and bilirubin) will be assessed before and after 30 h of paracetamol administration (T <0 and T = 30 h).

Venous blood samples are collected at the following times:

T = 0min, 15min, 30min, 45min, 60min, 90min, 120min, 180min, 240min, 300min, 360min, 24 hours, 24 hours 15min, 25 hours 30min, 27 hours and 30 hours.

VAMS VAMS samples are generated from the collected venous blood sample and from capillary blood obtained by a fingerstick. Only at T = 0 no VAMS are produced from capillary blood.

T = 30 min, 60 min, 120 min, 180 min, 360 min, 24h 15 min and 30 hours. (7 finger pricks)

In addition, the VAS pain score and Surgical Pleth index will also be monitored, as well as the consumption of piritramide via a patient-controlled intravenous analgesia pump (PCIA pump), to objectively evaluate pain relief in the current dosing regimen.

Visual Analog Scale and Surgical Pleth Index:

VAS pain scores are measured at rest and after movement (coughing) simultaneously with the SPI.

VAS T = 180min, 240min, 300min, 360min, 24h, 24h15, 25h30min, 27h and 30h SPI T = 180min, 240min, 300min, 360min, 24h, 24h15, 25h30min, 27h and 30h

Patients who are discharged within 24hrs and cannot complete the full measurement cycle are not considered dropouts.

statistical analysis

Fisher exact test for Categorical data. For continuous data with normal distribution: unpaired student t-test or rMANOVA for repeated measures. Mann-Whitney test as non-parametric test and to test the AUC 0-8hr for paracetamol + metabolites. The Wilcoxon rank test to test liver function samples. Acetaminophen and metabolite data are analyzed using non-linear mixed effects modelling NONMEM version 7.2. Bland- Altman and Passing & Bablok regression analysis for agreement between techniques.

F. significance

If this study reveals that 4g/day of paracetamol is insufficient to reach therapeutic plasma levels of paracetamol, then higher doses of paracetomol might be needed. If the results of the VAMS method are comparable to the venous blood samples, than future studies can use capillary samples to explore the concentrations of paracetamol and its toxic metabolites when higher doses of paracetamol are administered.

G. Flowchart

Inclusion criteria for obese patients:

* BMI> 35 kg.m-2 undergoing laparoscopic bariatric surgery.
* Patients >18 years old
* ASA physical classification II to III

Inclusion criteria for control patients:

* Patients 18.5 ≤ BMI ≤ 30 kg.m-2 undergoing elective laparoscopic surgery (Nissen procedure, inguinal hernia repair, laparoscopic bowel surgery and cholecystectomy).
* ASA physical classification I to III
* Patients > 18 yrs

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 < 70 years old (obese patients) Adult ≥ 18 years old (non-obese patients)
2. Able to comprehend, sign, and date the written informed consent document to participate in the clinical trial
3. Obese scheduled for laparoscopic bariatric surgery Non obese scheduled for laparoscopic surgery
4. Control group BMI ≥18.5 en <30 kg.m-2 or Obese group BMI > 35kg.m-2
5. ASA Class I, II or III as assigned by the anaesthesiologist

Exclusion Criteria:

1. Allergy or inability to tolerate "paracetamol"
2. Documented Liver disease or liver enzymes > 3X normal value
3. Kidney disease (eGFR < 30ml.min-1)
4. Participation in a clinical trial within the past 30 days
5. Chronic alcohol abuse or alcohol intake <72hrs
6. Gilbert-Meulengracht-syndroom
7. Chronic malnutrition
8. Intake of medication with influence on CYP2E1 or UDP-glucuronosyltransferase
9. Pregnancy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: control group is the cohort of patients with a BMI between 18,5 and 30 kg/m2. study group is the cohort of patients with a BMI over 35 kg/m2. All patients undergo laparscopic surgery because laparoscopy can affect liver function.
  since there are gender differences in acetaminophen metabolism, both cohorts were stratified into equal amounts of men and women.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
acetaminophen | first six hours after IV administration of the loading dose of 2g
  plasma concentrations and capillary blood concentrations
acetaminophen | the six hours after IV administration of the fifth dose of 1g acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen-glucuronide metabolite | the first six hours after IV administration of a loading dose of 2g acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen-glucuronide metabolite | the first six hours after IV administration of fifth dose of 1 g acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen-sulphate metabolite | the first six hours after IV administration of 2g IV acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen-sulphate metabolite | the six hours after IV administration of fifth dose of 1g IV acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen- Cysteine protein adduct | the first six hours after IV administration of 2 g loading dose of acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen- Cysteine protein adduct | the six hours after IV administration of the fifth dose of 1g acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen- mercapturate protein adduct | the first six hours after IV administration loading dose 2g acetaminophen
  plasma concentrations and capillary blood concentrations
acetaminophen- mercapturate protein adduct | the six hours after IV administration of the fifth dose of 1g acetaminophen
  plasma concentrations and capillary blood concentrations

SECONDARY OUTCOMES:
pain score using Visual analog scale at rest | hours after starting acetaminophen: 3,4,5,6, 24, 24:15, 25:30,27,30
  patient indicates the pain score on a visual analog scale ranging from 0-100mm
pain score using Visual analog scale after movement | hours after starting acetaminophen: 3,4,5,6, 24, 24:15, 25:30,27,30
  patient indicates the pain score on a visual analog scale ranging from 0-100mm
surgical pleth index (SPI) at rest | hours after starting acetaminophen: 3,4,5,6, 24, 24:15, 25:30,27,30
  non invasive measurement of the balance between nociception and antinociception ranging from 0-100.
surgical pleth index (SPI) after movement | hours after starting acetaminophen: 3,4,5,6, 24, 24:15, 25:30,27,30
  non invasive measurement of the balance between nociception and antinociception ranging from 0-100.
patient controlled intravenous analgesia: piritramide consumption | first 30 hours after starting acetaminophen or until discharge from the hospital
  piritramide consumption as a measure of the quality of pain relief with acetaminophen and ibuprofen.

CONTACTS AND LOCATIONS:
Overall Officials: Luc De Baerdemaeker, Md,PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Rongen A, Valitalo PAJ, Peeters MYM, Boerma D, Huisman FW, van Ramshorst B, van Dongen EPA, van den Anker JN, Knibbe CAJ. Morbidly Obese Patients Exhibit Increased CYP2E1-Mediated Oxidation of Acetaminophen. Clin Pharmacokinet. 2016 Jul;55(7):833-847. doi: 10.1007/s40262-015-0357-0. PMID 26818482